CLINICAL TRIAL: NCT00226902
Title: Integrated Studies in Vascular Reactivity and Anaemia Correction Therapy in Endstage Kidney Disease Patients
Brief Title: Vascular Reactivity in Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Interactedd
Record Dates: First submitted 2005-09-26; First posted 2005-09-27 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Failure, Chronic; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes; Hemoglobin; Dialysis; Vascular reactivity
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Changing hemoglobin concentration

SUMMARY:
Dialysis patients suffer from many problems with blood vessels and this is even more so for patients with the added complication of diabetes. Diabetics have a number of reasons for vascular disease and one of the new areas of research is looking at the cells that line the blood vessels, called endothelial cells. It is thought that the number of red blood cells in the blood (haemoglobin concentration) affects the function of these cells. There is very little information available on what haemoglobin level is best for dialysis patients. As diabetics account for almost 40% of dialysis patients worldwide it is important to understand the effect different haemoglobin levels will have on the blood vessels.

Hypothesis: Endothelial cell function and the related expansile capacity of blood vessels are affected by different haemoglobin concentrations [Hb] in dialysis patients.

DETAILED DESCRIPTION:
This project is going to ask dialysis patients (both diabetic and non-diabetic) to undergo a series of tests at three different time points over a one year period: a baseline set of tests, tested when haemoglobin is maintained at 130-140g/L and repeat the tests when haemoglobin is maintained at 105-115g/L. The current recommendation for haemoglobin is 110-120g/L. Patients will not be required to take any study medication but a specialist kidney doctor, using their usual medications of iron and erythropoietin therapy, will change their haemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years
2. Patients receiving either conventional haemodialysis 3-4 x week, for a duration of > 6 months or peritoneal dialysis for a duration >6 months
3. Stable dialysis access for at least 3 months (Permcath / PTFE / AVF)
4. On erythropoietin and iron therapy, with stable [Hb] x 2 months (105 - 135g/L)

Exclusion Criteria:

1. Uncontrolled BP: requiring dry weight or medication changes within 4 weeks prior to study
2. Patients with dysrhythmias
3. Pre dialysis SBP> 180 mmHg on > 2 times within a 2 week period
4. Between dialysis weight gain > 5% of body weight (if evident > 2 times/ 2 week period)
5. Soft tissue ulcers
6. Non traumatic amputations
7. Unstable cardiac function: ischaemic or non ischaemic events requiring modification of therapy, or admission to hospital within 3 months of study start: according to clinical discretion
8. Planned operative procedures within 6 months of study start (including Transplant, CABG, PTCA, vascular surgery)
9. Dementia
10. Clinical inability to comply with testing
11. Malignancy (active / under treatment)
12. Known hypo-responsiveness to ERT (>200U/kg/wk)
13. Evidence of chronic gastrointestinal bleeding
14. Inadequate dialysis (PRU < 65% or KT/V < 1.2)
15. Participation in investigational study within last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-09; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in pulse wave velocity at the three different haemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P McMahon, MD, Principal Investigator — Melbourne Health
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia